CLINICAL TRIAL: NCT03645083
Title: Improving Treatment Adherence in Acupuncture Patients: A Randomized Controlled Trail
Brief Title: Patient Adherence to Acupuncture Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, David Black, Assistant Professor of Preventive Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-17-00008
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Adherence, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telephone call (Experimental): Participants receive a telephone call reminder three days after their initial visit
  Interventions: Behavioral: Telephone call
- Text message (Experimental): Participants receive a text message reminder three days after their initial visit
  Interventions: Behavioral: Text message
- Control (No Intervention): Participants do not receive any intervention after their initial visit

INTERVENTIONS:
Behavioral: Telephone call — Participants in the intervention group receive a one-time telephone call reminder to attend follow-up treatment at the acupuncture clinic
  Arms: Telephone call
Behavioral: Text message — Participants in the intervention group receive a one-time text messaging reminder to attend follow-up treatment at the acupuncture clinic
  Arms: Text message

SUMMARY:
Adherence to treatment recommendation remains low among acupuncture patients. This study aims to examine whether implementing a post-initial visit follow-up strategy can improve adherence rate. Adult patients visiting the acupuncture clinic for a new treatment will be randomized to receive a telephone call or a text-message three days after their initial visit against a control group. We will enroll up to 160 participants between February and December 2017, to ensure we can reach 120 subjects in the analysis who completed the baseline survey. Participants recruitment will take place at the Emperor's College of Traditional Oriental Medicine Acupuncture Clinic. Assessments will be conducted via surveys at four times points, Day 0 (date of enrollment), Day 3, Day 10 and Day 30. Additional data will also be collected via chart review. Primary outcome will be assessing whether participants return for any follow-up visit within 30 days after the initial treatment. Secondary outcomes will examine if factors such as expectations, intention, satisfaction, and potential barriers would predict the primary outcome.

DETAILED DESCRIPTION:
This randomized controlled trial will deliver two interventions: (1) telephone call reminder and (2) text messaging reminder.

Participants who meet study eligibility criteria based on intake assessment will be recruited and complete baseline assessment immediately after they receive acupuncture treatment. There will be 40 participants in each of the two intervention groups and the no intervention control group.

Participants will be adults who visit the Emperor's College Acupuncture Clinic for a new treatment consultation on the date of the enrollment.

The telephone call and text messaging intervention is a one-time reminder system delivered to the participants based on the study random assignment, three days after the initial visit. A research assistant will be contacting the participants based on the assigned interventions.

There are three data collection points, 1) baseline (during initial visit), 2) 10 days after the initial visit, and 3) 30 days after the initial visit. Data will be collected via a tablet (baseline) and online survey (Day 10 and Day 30) through a secure online survey platform. Baseline assessment will occur prior to randomization, and post-intervention assessments will occur at 10 to 30 days after the initial visit.

Number of follow-up treatments for the same health concern will be collected for all enrolled participants from the participants' clinical record.

ELIGIBILITY:
Inclusion Criteria:

* Outside patients seeking acupuncture treatment at Emperor's College Clinic
* Age 18 and above
* English-speaking
* Starting a new treatment at the day of recruitment
* Own a mobile device
* Mobile device has text-messaging capability
* Visiting the Master's Clinic at Emperor's College

Exclusion Criteria:

* Emperor's College's students or staffs seeking acupuncture treatment
* Patients visiting the faculty observation theater, ear acupuncture clinic and private clinic
* Patients returning for a follow-up acupuncture visit at the day of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Attendance to follow-up treatment | Within 30 days after participants' initial visit
  Participants attending acupuncture follow-up treatments

SECONDARY OUTCOMES:
Total number of follow-up treatments | Within 30 days after participants' initial visit
  The total number of follow-up treatments by participants

CONTACTS AND LOCATIONS:
Overall Officials: David Black, PhD, Study Director — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD